CLINICAL TRIAL: NCT00127257
Title: Biofeedback for Fecal Incontinence and Constipation
Brief Title: Biofeedback for Dyssynergic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RO1 DK57048b (completed); R01DK057048 (NIH)
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Constipation
Keywords: Constipation; Biofeedback; Dyssynergia; Pelvic floor dyssynergia; Outlet dysfunction
MeSH Terms: conditions — Constipation; Ataxia | interventions — Biofeedback, Psychology; Diazepam

INTERVENTIONS:
Behavioral: Biofeedback
Drug: Diazepam
Behavioral: Pelvic floor retraining

SUMMARY:
Constipation affects 4% of adults in the United States (U.S.). An estimated half of constipated patients are unable to relax pelvic floor muscles during defecation, a type of constipation called pelvic floor dyssynergia (PFD). Biofeedback has been recommended for the treatment of constipation because uncontrolled studies over the past 10 years suggest that these treatments are as effective as medical or surgical management and involve no risk. However, placebo-controlled trials are still lacking. The aims of this study are:

* to compare biofeedback to alternative therapies for which patients have a similar expectation of benefit;
* to identify which patients are most likely to benefit; and
* to assess the impact of treatment on quality of life.

DETAILED DESCRIPTION:
This study is a long-term prospective, single-blind study comparing biofeedback for pelvic floor dyssynergia to a skeletal muscle relaxant drug (diazepam 5 mg two hours before attempted defecation) and to placebo medication. Prior to randomization, patients will first receive medical therapy (laxatives and education) for 4 weeks and only those remaining constipated will be randomized. Physiological tests of anal canal pressure during straining to defecate and ability to pass a 50-ml air filled balloon will be tested before and after treatment. Patients will keep a diary throughout baseline and treatment, and they will be reassessed at 3, 6, and 12 months follow-up. Treatment will consist of 6 clinic visits at 2-week intervals. The investigators will develop a detailed treatment manual for this disorder which would permit other investigators to replicate their study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 16 or above who have symptoms of constipation due to pelvic floor dyssynergia

Exclusion Criteria:

* Pregnancy (because of the possibility of randomization into the diazepam group)
* Prior history of biofeedback treatment for pelvic floor disorders

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117
Dates: Start 1999-09; Study Completion 2006-06

PRIMARY OUTCOMES:
Proportion of subjects reporting adequate relief per treatment group

SECONDARY OUTCOMES:
Demonstrate association of improvement in quality of life with treatment outcome
Identify predictors of successful treatment outcome
Describe physiological mechanism of treatment effects

CONTACTS AND LOCATIONS:
Overall Officials: William E Whitehead, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Department of Medicine, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Palsson OS, Heymen S, Whitehead WE. Biofeedback treatment for functional anorectal disorders: a comprehensive efficacy review. Appl Psychophysiol Biofeedback. 2004 Sep;29(3):153-74. doi: 10.1023/b:apbi.0000039055.18609.64. PMID 15497616
- [Background] Heymen S, Jones KR, Scarlett Y, Whitehead WE. Biofeedback treatment of constipation: a critical review. Dis Colon Rectum. 2003 Sep;46(9):1208-17. doi: 10.1007/s10350-004-6717-8. PMID 12972965
- [Background] Whitehead WE, Heymen S, Schuster MM. Motility as a therapeutic modality: biofeedback treatment of gastrointestinal disorders. Chapter 27. In MM Schuster, MD Crowell, KL Koch (Eds.), Schuster Atlas of Gastrointestinal Motility in Health and Disease. London, BC Decker Inc. 2002; 381-397.
- [Background] Heymen S, Jones KR, Ringel Y, Scarlett Y, Drossman D, Whitehead WE (abstract). Biofeedback for fecal incontinence and constipation: the role of medical management and education. Gastro 2001 (suppl 1):120, A397.
- [Result] Heymen S, Scarlett Y, Whitehead WE. Constipated subjects reporting physical abuse are more likely to fail an education/medical management intervention. Am J Gastroenterol Suppl 2004;99:T1364
- [Result] Heymen S, Scarlett Y, Whitehead WE. Severity of constipation and anxiety predict failure to improve with conservative medical treatment for constipation. Am J Gastroenterol Suppl 2004;99:T1370
- [Result] Heymen S, Scarlett Y, and Whitehead WE. Elevated Beck Depression Inventory (BDI) Scores Predict Biofeedback Treatment Failure for Fecal Incontinence and Constipation (abstract). Gastroenterology 2003,124:4(suppl 1)A-685.